CLINICAL TRIAL: NCT02472860
Title: Feasibility and Effectiveness of Computerized Cognitive Training in Adolescents With Autism Spectrum Disorder
Acronym: MGHTCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Deborah Munroe Noonan Memorial Research Fund (Other)
Responsible Party: Principal Investigator, Alysa Emily Doyle, PhD, Assistant Professor of Psychiatry, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2015P000610
Record Dates: First submitted 2015-06-08; First posted 2015-06-16 (Estimated); Last update posted 2018-03-27 (Actual); Status verified 2018-03

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism Spectrum Disorder; Neuroplasticity-based Cognitive Training
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive Training (Experimental): Targeted Cognitive Training (TCT)
  Interventions: Behavioral: Targeted Cognitive Training (TCT)
- Control Condition (Placebo Comparator): Youth appropriate online games
  Interventions: Other: Youth Appropriate Online Games

INTERVENTIONS:
Behavioral: Targeted Cognitive Training (TCT) — The investigators have selected a set of computer exercises designed to specifically target aspects of cognition relevant to autism spectrum disorder (including attention and executive functions). The tasks were designed to benefit subjects through principles of learning dependent plasticity.
  Arms: Cognitive Training
Other: Youth Appropriate Online Games — Engaging games not designed to improve cognition
  Arms: Control Condition

SUMMARY:
The investigators will conduct a randomized placebo-controlled trial of a computerized intervention targeting cognition in 30 teens with autism spectrum disorder.

DETAILED DESCRIPTION:
Given the limited options for treatments to improve the core symptoms of autism spectrum disorder (ASD), strategies that could target secondary features of the condition and improve quality of life for affected individuals are critical. Neuroplasticity-based cognitive training has been found to improve cognition in youth with attention deficit hyperactivity disorder (ADHD) and in adults with schizophrenia. In this trial, the investigators are seeking to extend the relevance of computerized cognitive training to youth with ASD. Given the literature, the investigators hypothesize that computerized cognitive training will produce gains in untrained cognitive tasks and behavioral ratings of executive functions in youth with ASD. The investigators will assess aspects of attention and executive functions in 30 affected youth and randomize them 1:1 to either neuroplasticity based cognitive tests or enjoyable age-appropriate computer games not intended to improve cognition. Cognition will be assessed again after 15 hours of training over 6 weeks and then again at a three month follow up.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnostic and Statistical Manual of Mental Disorders (DSM)-5 ASD or previously diagnosed DSM-IV autistic disorder, Asperger's disorder or pervasive developmental disorder not otherwise specified (NOS) and who continue to manifest symptoms in core domains
2. Current ASD symptomatology at time of enrollment
3. Evidence of decrements in at least one of three target cognitive domains (mental flexibility/abstraction, working memory, or attention).

Exclusion Criteria:

1. Intellectual Disability
2. A known comorbid neurodevelopmental disorder with possible association with autism (i.e., fragile X syndrome, tuberous sclerosis, Angelman syndrome, Prader-Willi syndrome, Williams syndrome, neurofibromatosis, mitochondrial disorder).
3. Nonverbal or minimal verbal ability
4. No computer/internet connection at home
5. No family member with e-mail
6. Patients likely to have a change in therapeutic treatments within the next 6 weeks

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 29 (Actual)
Dates: Start 2015-06; Primary Completion 2017-08-02 (Actual); Study Completion 2017-08-02 (Actual)

PRIMARY OUTCOMES:
Cambridge Neuropsychological Test Automated Battery (CANTAB) | 6 weeks
  Computerized test

CONTACTS AND LOCATIONS:
Overall Officials: Alysa E Doyle, PhD, Principal Investigator — Massachusetts General Hospital